CLINICAL TRIAL: NCT03941717
Title: A Randomized Controlled Trial Testing the Effectiveness of a Mindfulness-Based Intervention for Both Parents and Children During Child Venipuncture
Brief Title: Testing the Effectiveness of a Parent and Child Mindfulness-Based Intervention for Child Venipuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Principal Investigator, Meghan McMurtry, Associate Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REB 5481
Record Dates: First submitted 2019-05-05; First posted 2019-05-08 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Pain; Needle Stick
Keywords: pain management; children; parents; mindfulness
MeSH Terms: conditions — Pain; Needlestick Injuries; Agnosia

STUDY DESIGN:
Intervention Model Description: The study will be a single-site, two-arm, parallel group RCT with an intervention group (mindfulness-based intervention) and control group (unfocused-attention task, no active components).
Who Masked: Participant
Masking Description: Participants will not be made explicitly aware of which group (intervention or control) that they have been allocated. Participants in each group will be provided with a tablet and guided through an audio activity. Further, participants will not be made aware of the kind of intervention being used, however, it is possible that participants may become aware of the nature of their treatment allocation in the mindfulness group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Condition (Experimental): Parents and children in the mindfulness intervention condition will be provided with a tablet and accompanying headphones, and will listen to pre-recorded audio of a mindfulness activity. There is a parent and child version of the mindfulness intervention. Both scripts were developed by Siegel and Bryson (2011), and include a parent and child version of a mindfulness activity targeting worries and anxiety. Adjustments to the child script were informed by the work of Petter and colleagues (2013). Adjustments to the parent script were informed by the work of Garland and colleagues (2015). This activity will last 5-minutes.
  Interventions: Other: Mindfulness-Based Condition
- Unfocused attention Condition (Sham Comparator): Parents and children in the unfocused attention condition will be provided with a tablet and accompanying headphones, and will listen to pre-recorded audio of an unfocused attention activity. There is a parent and child version of this activity. The parent version has been validated in other research with healthy adults as a control for a mindfulness intervention (Garland, Hanley, Farb, & Froeliger, 2015). This script was condensed in time from the original reading. The child version of the activity was developed for the current study, and was adapted from a mind-wandering script used for children aged 7-12 in past research (Spann, 2016). It was also informed by the unfocused attention script used for parents (Garland, Hanley, Farb, & Froeliger, 2015), and work by Cahn and Polich (2009). This activity will last 5-mintues.
  Interventions: Other: Unfocused attention Condition

INTERVENTIONS:
Other: Mindfulness-Based Condition — Each script for the mindfulness-based intervention was slightly modified to fit the context of a venipuncture, and begins with instructions to take deep breaths. Both scripts aim to cultivate present moment awareness of experiences, curiosity, nonjudgement, and acceptance of experiences as they unfold. In particular, the scripts ask that the participant visualize their worries and feelings as a cloud in the sky, and probes for curious thoughts about these experiences. The temporary nature of sensations is described, and the participant is asked to keep this openness and curiosity during the venipuncture.
  Arms: Mindfulness-Based Condition
Other: Unfocused attention Condition — Each script for the unfocused attention task instructs participants to allow their mind and thoughts to roam. The aim is to encourage the participant to continue thinking and mind wandering as they typically would.
  Arms: Unfocused attention Condition

SUMMARY:
This study investigates the impact of mindfulness-based intervention for children undergoing a blood-draw and their accompanying parent on (a) child ratings of pain and fear, (b) parent and child ratings of parent distress, and (c) parent perceptions of child pain and fear. Half of the parent-child pairs will receive the mindfulness-based intervention, while half will receive an unfocused-attention task to serve as a comparison with no active component.

DETAILED DESCRIPTION:
To date, there are no randomized controlled trials (RCT) involving a mindfulness intervention for pediatric acute pain. Moreover, this will be the first study to investigate a parent mindfulness intervention in the context of child acute pain. Within a randomized control trial, the objectives of this study are to test the effectiveness of a mindfulness-based intervention for children undergoing a venipuncture and their accompanying parent on (a) child ratings of pain and fear, (b) parent and child ratings of parent distress, and (c) parent perceptions of child pain and fear. Participants will complete questionnaires immediately before and after child venipuncture. This study aims to offer a novel intervention that may improve both parent and child experience during a stressful situation in which parent and child unmanaged distress has deleterious effects. The long-term objectives of this line of research are to improve extant pain management interventions for children undergoing needle-pokes or other painful procedures.

Moderator Aims: To identify possible moderators of a differential treatment outcome (parent and child responses during the needle-poke). These psychological factors include parent and child state catastrophizing, trait experiential avoidance, and trait mindfulness which will be investigated as moderators of the impact of experimental group on the primary outcomes of child self-reported pain and fear, and secondary outcome of parent self-reported distress.

ELIGIBILITY:
Inclusion Criteria:

* Proficiency in English

Exclusion Criteria:

* Major developmental delays in child

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Child pain during the needle: Numeric Rating Scale (NRS) | Within two minutes following the needle-poke.
  Between group changes in child self-reported pain as rated on a Numeric Rating Scale (NRS). The NRS has been used to assess pain intensity in children aged 7 and older during acutely painful procedures (Hsieh et al., 2017; Pagé, Stinson, Campbell, Isaac, & Katz, 2013; Vervoort et al., 2011).The NRS is rated on an 11-point numerical rating scale, ranging from 0 ("no pain") to 10 ("a lot of pain").
Child fear during the needle | Within two minutes following the needle-poke.
  Between group changes in child self-reported fear as rated on a Numeric Rating Scale (NRS). The NRS has been used to assess child fear in children aged 7 and older during acutely painful procedures (Hsieh et al., 2017; Vervoort et al., 2011). The NRS is rated on an 11-point numerical rating scale, ranging from 0 ("not scared") to 10 ("very scared").

SECONDARY OUTCOMES:
Child perceptions of parent distress | Within five minutes following the needle-poke.
  Between group changes in child perceptions of parent fear as rated on a NRS (researcher generated). Children will be asked to "Tell us how upset you think your parent was during the needle". This item will be rated on an 11-point numerical rating scale, ranging from 0 ("not at all") to 10 ("extremely").
Parent distress | Within five minutes following the needle-poke.
  Between group changes in parent self-report distress as rated on a NRS. Parents will be asked to provide ratings indicating their level of distress experienced on a NRS (researcher generated). For the purpose of the current study, the NRS will ask parents to "Tell us how distressed you were during the needle". The NRS is rated on an 11-point numerical rating scale, ranging from 0 ("not at all") to 10 ("extremely").

OTHER OUTCOMES:
Parent perceptions of child pain | Within five minutes following the needle-poke.
  Between group changes in parent report of child pain as rated on a NRS (Vervoort et al., 2011). Parents will be prompted to provide ratings corresponding to how much pain they think their child experienced. The NRS is rated on an 11-point numerical rating scale, ranging from 0 ("no pain") to 10 ("a lot of pain").
Parent perceptions of child fear | Within five minutes following the needle-poke.
  Between group changes in parent report of child fear as rated on a NRS (Vervoort et al., 2011). Parents will be prompted to provide ratings corresponding to how much pain they think their child experienced. The NRS is rated on an 11-point numerical rating scale, ranging from 0 ("not scared") to 10 ("very scared").

CONTACTS AND LOCATIONS:
Overall Officials: C. Meghan McMurtry, PhD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsieh LY, Chen YR, Lu MC. Efficacy of cold application on pain during chest tube removal: a randomized controlled trial: A CONSORT-compliant article. Medicine (Baltimore). 2017 Nov;96(46):e8642. doi: 10.1097/MD.0000000000008642. PMID 29145288
- [Background] Page MG, Stinson J, Campbell F, Isaac L, Katz J. Identification of pain-related psychological risk factors for the development and maintenance of pediatric chronic postsurgical pain. J Pain Res. 2013;6:167-80. doi: 10.2147/JPR.S40846. Epub 2013 Mar 5. PMID 23503375
- [Background] Vervoort T, Goubert L, Vandenbossche H, Van Aken S, Matthys D, Crombez G. Child's and parents' catastrophizing about pain is associated with procedural fear in children: a study in children with diabetes and their mothers. Psychol Rep. 2011 Dec;109(3):879-95. doi: 10.2466/07.15.16.21.PR0.109.6.879-895. PMID 22420118
- [Background] Spann, C. A. (2016). Mindfulness and mind-wandering: the impact of brief interventions on child affect, arousal, and cognition. The University of Texas at Arlington. Retrieved from https://uta-ir.tdl.org/uta-ir/bitstream/handle/10106/25806/SPANN-DISSERTATION-2016.pdf?sequence=1&isAllowed=y
- [Background] Cahn BR, Polich J. Meditation (Vipassana) and the P3a event-related brain potential. Int J Psychophysiol. 2009 Apr;72(1):51-60. doi: 10.1016/j.ijpsycho.2008.03.013. Epub 2008 Sep 23. PMID 18845193
- [Background] Garland EL, Hanley A, Farb NA, Froeliger BE. State Mindfulness During Meditation Predicts Enhanced Cognitive Reappraisal. Mindfulness (N Y). 2015 Apr 1;6(2):234-242. doi: 10.1007/s12671-013-0250-6. PMID 26085851
- [Background] Petter M, Chambers CT, MacLaren Chorney J. The effects of mindfulness-based attention on cold pressor pain in children. Pain Res Manag. 2013 Jan-Feb;18(1):39-45. doi: 10.1155/2013/857045. PMID 23457685
- [Background] Siegel, D. J., & Bryson, T. P. (2011). The whole-brain child : 12 revolutionary strategies to nurture your child's developing mind. Delacorte Press. Retrieved from https://books.google.ca/books/about/The_Whole_Brain_Child.html?id=APzgCL8mgHUC&printsec=frontcover&source=kp_read_button&redir_esc=y#v=onepage&q&f=false
- [Derived] Constantin KL, Moline RL, Pillai Riddell R, Spence JR, Fiacconi CM, Lupo-Flewelling K, McMurtry CM. Parent and child self- and co-regulation during pediatric venipuncture: Exploring heart rate variability and the effects of a mindfulness intervention. Dev Psychobiol. 2022 Jul;64(5):e22277. doi: 10.1002/dev.22277. PMID 35603416